CLINICAL TRIAL: NCT00515541
Title: Effect of the Omega n3 Fatty on Human Platelet Function
Brief Title: Lovaza's Effect on the Activation of Platelets
Acronym: LEAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Invitrox (Industry)
Collaborators: Reliant Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-1068
Record Dates: First submitted 2007-08-10; First posted 2007-08-13 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-06

CONDITIONS: Cardiovascular Disease; Bleeding
Keywords: Platelet; Cardiovascular; Lipid; Fish Oil; Omega 3; DHA; EPA; Bleeding; Clotting; platelet function; Lipid profile; Weight and Bleeding risk
MeSH Terms: conditions — Cardiovascular Diseases; Hemorrhage; Thrombosis; Body Weight | interventions — Omacor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A (Active Comparator): Patient is not on Aspirin, Clopidogrel, or Warfarin and is taking escalating doses of study drug.
  Interventions: Drug: Lovaza
- B (Active Comparator): Patient is on regular dose of Aspirin ( < or = 325mg). Patient is not taking Clopidogrel or Warfarin and is taking the escalating doses of Lovaza
  Interventions: Drug: Lovaza
- C (Active Comparator): Patient is taking regularly 75mg of clopidogrel daily and Aspirin (< or = 325mg) and not taking Warfarin and is taking the escalating doses of Lovaza
  Interventions: Drug: Lovaza
- D (Active Comparator): Patient is regularly taking Warfarin daily and Aspirin (< or = 325mg)and is not taking Clopidogrel and is taking the escalating doses of Lovaza
  Interventions: Drug: Lovaza

INTERVENTIONS:
Drug: Lovaza — First 6 weeks period take 1 gram Lovaza capsule daily 2nd 6 weeks period take 2 grams of Lovaza (2 1 gram capsules) daily 3rd 6 weeks period take 4 grams of Lovaza (4 1 gram capsules) daily 4th 6 weeks period take 8 grams of Lovaza (8 1 gram capsules) daily

SUMMARY:
This study is to determine the effects of Lovaza in platelet function studies

DETAILED DESCRIPTION:
Cardiovascular disease remains a leading cause of death in North America (1). Uncontrolled platelet activation, adhesion and aggregation initiated by vessel wall plaque rupture are thought to be responsible for acute vascular occlusion in many situations (2-5). Although many platelet inhibition drugs are available, all currently available drugs have undesirable toxicity profiles (6-8). Thus, reduction in toxicity and improved management of patients with thrombotic diseases remains an unmet medical need.

Platelet activation plays a pivotal role in the pathogenesis of acute coronary syndromes, strokes and other thrombophilic diseases. Atheromatous plaque rupture changes the shear forces of blood flowing over the injured vessel surface and also exposes collagen as well as other prothrombotic factors (9-11). As the initial hemostatic event, platelets become activated and cover the injured surface. Following platelet activation highly active substances like adenosine diphosphate (ADP) and thromboxane A2 (TxA2) are released from the platelet to promote and recruit further platelet aggregation to the injury site (12). If this process proceeds unabated, as it often does in atherosclerotic diseases, the vessel becomes occluded and infarction may follow.

Lovaza® (Reliant Pharmaceutical Inc., Liberty Corner, NJ), a commercially available formulation that contains 90 % omega-3-acid ethyl esters (46% eicosapentaenoic acid -EPA- and 38% docosohexaenoic acid -DHA-), has the potential ability to modify the recruitment of additional platelets to the growing thrombus by promoting synthesis of thromboxane A3 (TxA3), a poor platelet activator, instead of thromboxane A2, a potent platelet activator. Agents used to inhibit platelet function such as aspirin and clopidogrel are not always effective (13-16). Unfortunately, some patients do not respond to these therapeutics (17-24). Realistic numbers for patient resistance to these drugs are probably 10-15% for ASA and 20-30% for clopidogrel. Almost all resistant patients have less favorable outcomes and are unaware of this potentially life-threatening problem until a severe cardiac adverse event occurs. Lovaza® may add additional therapeutic benefit to these patients.(25,26) Beyond the occasional patient with complaints of eructation or a "fishy" taste in their mouth, Lovaza® has a benign toxicity profile. If Lovaza® can be shown to have a clinically relevant anti-platelet effect, it may have a use to either replace or reduce the dose of more toxic anti-platelet agents.

The proposed biochemical mechanism for the anti-platelet effect of omega n3 fatty acids is based on modifications in platelet prostaglandin metabolism (27-31). Cellular membranes are primarily composed of phospholipids (PL). The backbone of PL's is glycerol. The glycerol hydroxyl groups in position 1 and 2 bind two fatty acid molecules through formation of ester bonds (31). The third hydroxyl binds the so-called head group, which may be choline, inositol, ethanolamine or serine. At least in the case of platelets the fatty acid at the C-2 position is often the unsaturated arachidonic fatty acid (an omega n6 fatty acid). When Lovaza® is ingested (an omega n3 fatty acid), the unsaturated fatty acid at the C2 position can be DHA or EPA. Several important differences result from this substitution including an important effect on platelet function. As part of the platelet activation process, phospholipase A2 clips the fatty acid at the C-2 position, either arachidonic acid or DHA/EPA (31). In the case of the platelet, the fatty acid is then metabolized through an enzyme called COX-1 to a thromboxane (32-35). When the fatty acid is arachidonic acid, thromboxane A2 is synthesized (TxA2). TxA2 is a very potent platelet activator and vasoconstrictor. In the case of DHA or EPA, a series 3 TxA3 is synthesized, a poor platelet activator and vasoconstrictor (32-35). Production of TxA3 underlies the potential anti-platelet effect of Lovaza®.

The second effect of DHA inclusion in PL's is a newly discovered alteration in the cell membrane structure. It is now well established that DHA promotes "lipid raft" formation in cellular membranes (36-38). These rafts, primarily composed of sphingomyelin and cholesterol, form the sites where some transmembrane proteins can be inserted into the membrane. These transmembrane proteins may be sites for ion channels or receptors that define important cellular functions and can be a means to activate cells. Thus, DHA's ability to promote raft formation may have a profound beneficial effect on platelet function.

Since it is the Lovaza®-alteration of the platelet membrane that leads to its clinical benefit, assays to determine how the lipid composition of the platelet membrane changes after ingestion of Lovaza® will be carried out. The concept of these experiments is fairly simple. A standard well-established 1H NMR method will be used to detect changes in the lipid composition of the platelet membrane as a function of the Lovaza® dose (39-41). From these experiments we will be able to prove that DHA or EPA from Lovaza® is actually directly incorporated into a platelet membrane

ELIGIBILITY:
Inclusion Criteria:

* Males or females older than 18 years old who are able to ingest omega n3 fatty acids are eligible for this trial and are:
* On no antiplatelet and anticoagulation therapy, OR
* On chronic therapy with warfarin or aspirin alone (< or =325 mg/day)or combination therapy with clopidogrel and aspirin (< or =325 mg/day).
* The subject must be able to read, understand, and sign an informed consent form and follow protocol.
* To be enrolled in the study, subjects must be clinically stable on stable medical therapy throughout the duration of the study and meet the following criteria:
* Healthy volunteers
* Volunteers with stable coronary artery disease are those with:
* Prior MI (>1 month) OR
* Prior revascularization: angioplasty ± stenting (> 1 month) OR
* Coronary artery bypass grafting (>3 months) OR
* Documented disease on coronary angiography.
* No planned no planned procedures or changes in medical therapies over the 24-week duration of the study
* Volunteers with stable atrial fibrillation are those with:
* Rate-controlled or paroxysmal atrial fibrillation on stable antiarrhythmic therapy.
* On a stable dose of warfarin and regular follow-up in an anticoagulation ("coumadin") clinic.
* No planned changes in antiarrhythmic therapies or cardioversion during the duration of the study.
* No recent admissions for atrial fibrillation (> 3 months)
* Subjects may not ingest other drugs known to cause a significant platelet abnormality while participating in this trial. (See list of prohibited medications, as outlined in Section 9)
* Patients must be assessable to the investigator for scheduled clinic visits during the duration of the trial.
* All female subjects of child bearing potential must have a negative serum pregnancy test prior to randomization and not plan on getting pregnant for the duration of the study.

Exclusion Criteria:

* Any medical condition that would preclude ingestion of omega n3 fatty acids (Lovaza®).
* Subjects taking nutritional supplements of fish oil or flaxseed oil. These patients may become eligible if they are willing to discontinue these nutritional supplements for a 2-week washout period.
* Any other medical condition that would adversely affect the study objectives.
* Chronic medical conditions known to be associated with abnormal platelet function including:
* Liver dysfunction including abnormal liver function tests (AST, ALT, or alkaline phosphatase > upper limit of normal), known cirrhosis or chronic hepatitis.
* Chronic kidney disease with a calculated creatinine clearance < 60 ml/min (MDRD) and/or a serum creatinine > 2.0 mg/dl.
* History of significant anemia, or baseline hemoglobin < 11.0 g/dl.
* Baseline PT>ULN, INR>1.3, and aPTT>ULN in subjects who are not on chronic warfarin therapy.
* History of thrombocytopenia, or baseline platelet count of < 100,000
* History of thrombocytosis, or baseline platelet count of > 600,000
* Known bleeding diathesis and/or congenital hemostasis disorder and/or congenital platelet abnormalities.
* Any history of stroke in the past 12 months.
* History of peptic ulcer disease in the past year or gastrointestinal bleeding in the last 3 months.
* Genitourinary bleeding in the last 3 months.
* HIV or other infectious diseases that would expose laboratory personnel to unacceptable risks.
* Treatment within 30 days with an antiplatelet agent other than aspirin or clopidogrel such as eptifibatide, tirofiban or abciximab.
* Treatment within the past 7 days with unfractionated or low-molecular- weight heparin.
* Allergy to iodine, fish, or other components of the study drug.
* Alcohol or substance abuse.
* Emotionally or psychiatrically unstable.
* Use of any investigational drug or device within the past 30 days
* Any other factor that the investigator feels would put the patient at increased risk if participating in the study.
* Any Terminal illness or illness that may cause mortality that could obscure the results of the test in any way for them to appear inaccurate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauricio Cohen, MD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Result] Cohen MG, Rossi JS, Garbarino J, Bowling R, Motsinger-Reif AA, Schuler C, Dupont AG, Gabriel D. Insights into the inhibition of platelet activation by omega-3 polyunsaturated fatty acids: beyond aspirin and clopidogrel. Thromb Res. 2011 Oct;128(4):335-40. doi: 10.1016/j.thromres.2011.04.023. Epub 2011 May 28. PMID 21621252

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at the Carolina Center for Clinical Trials at the University of North Carolina at Chapel Hill campus. Enrollment period: 9/24/07 through 10/13/08.
Groups:
- Group A: Subjects on Lovaza Only: Group A: Subject is healthly and not on Aspirin, Clopidogrel, or Warfarin. Subjects will be taking escalating doses of the study drug (Lovaza)up to 24 weeks.
- Group B: Subjects on Lovaza Plus Aspirin: Group B: Subject is only taking Aspirin (< or = 325mg) daily. Subjects will be taking escalating doses of study drug (Lovaza) in addition to aspirin up to 24 weeks.
- Group C: Subjects on Lovaza Plus Clopidogrel and Aspirin: Subject is regularly taking Clopidogrel (75mg)and Aspirin (< or = 325mg)daily, and not taking Warfarin. Subjects will be taking escalating doses of study drug (Lovaza)in addition to Clopidogrel and Aspirin up to 24 weeks.
- Group D: Subjects on Lovaza Plus Warfarin and Aspirin: Subject is regularly taking Warfarin and Aspirin (< or = 325mg)daily, and not taking Clopidogrel. Subjects will be taking escalating doses of study drug (Lovaza)in addition to Warfarin and Aspirin up to 24 weeks.
Period: Overall Study
Arm/Group | Group A: Subjects on Lovaza Only | Group B: Subjects on Lovaza Plus Aspirin | Group C: Subjects on Lovaza Plus Clopidogrel and Aspirin | Group D: Subjects on Lovaza Plus Warfarin and Aspirin
Started | 10 | 12 | 10 | 11
6 Weeks (1 gm Lovaza) | 10 | 10 (One subject pulled after baseline. One subject pulled due to no show for appt.after baseline) | 10 | 10 (One subject pulled due to no show for appt. after baseline.)
12 Weeks (2 gm Lovaza) | 10 | 10 | 10 | 10
18 Weeks (4 gm Lovaza) | 10 | 9 (One subject withdrew at 12 weeks due to acquired bleeding disorder present before enrolling.) | 10 | 9 (One subject withdrew at 14 weeks with GI problems.)
24 Weeks (8 gm Lovaza) | 10 | 7 (Two subjects withdrew at 20 and 21 weeks due to nausea. Subjects were closed out early.) | 10 | 6 (Three subjects withdrew after 18 weeks (1 GI problem, 1 undefined medical problem, 1 no show))
Completed | 10 (All subjects completed 24 weeks.) | 7 | 10 (All subjects completed 24 weeks.) | 6
Not Completed | 0 | 5 | 0 | 5
Not completed — Physician Decision | 0 | 2 | 0 | 1
Not completed — No show for appointments | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Population: The number of subjects for baseline does not represent the number of subjects that completed the 24 week study.
Groups:
- Group A: Subject on Lovaza Only: Group A: Subject is not on Aspirin, Clopidogrel, or Warfarin. Subject is taking escalating doses of study drug (Lovaza)over a 24 week period.
- Group. B: Subject on Lovaza + Aspirin: Group B: Subject on Aspirin (< or = 325mg and is not taking Clopidogrel or Warfarin. Subject is taking escalating doses of Lovaza over a 24 week period.
- Group C: Subject on Lovaza + Clopidogrel + Aspirin: Group C: Subject is taking Clopidogrel 75mg)and Aspirin (< or = 325mg) and not taking Warfarin. Subject is taking escalating doses of Lovaza over a 24 week period.
- Group D: Subject on Lovaza + Warfarin + Aspirin: Group D: Subject is taking Warfarin and Aspirin (< or = 325mg)and is not taking Clopidogrel. Subject is taking escalating doses of Lovaza over a 24 week period.
- Total: Total of all reporting groups
Arm/Group | Group A: Subject on Lovaza Only | Group. B: Subject on Lovaza + Aspirin | Group C: Subject on Lovaza + Clopidogrel + Aspirin | Group D: Subject on Lovaza + Warfarin + Aspirin | Total
Number analyzed (Participants) | 10 | 12 | 10 | 11 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 12 | 10 | 11 | 43
  >=65 years | 0 | 0 | 0 | 0 | 0
Gender [Number; unit: participants]
  Female | 3 | 4 | 5 | NA — The reporting site did not supply this information to Invitrox. We have requested information but have been informed that it is not available.Group D was not included in final report. | 12
  Male | 7 | 8 | 5 | NA — The reporting site did not supply this information to Invitrox. We have requested information but have been informed that it is not available.Group D was not included in final report. | 20
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 10 | 11 | 43

OUTCOME MEASURES:

1. Primary Outcome: Platelet Aggegation (Arachiodonic Acid)Using a PAP-8E (BioData Corp.)
Description: The PAP-8E measures platelet aggregation in platelet rich plasma (PRP). Platelet responses to a series of common agonists cause changes in optical density that are measured. The instrument is blanked (100% baseline (optimal transmission)) by inserting a platelet poor plasma (PPP) specimen into the appropriate channel. The PRP is then inserted into the same well. The difference in optical density between the PPP and the PRP 0% baseline (optical transmission) is recorded for several minutes when the agonist reagent is added to the PRP.
Time Frame: up to and including closeout at 24 weeks
Population: Based on number of subjects completing 24 weeks
Measure: Median (Inter-Quartile Range); unit: percent
Groups:
- Group A: Subject on Lovaza Only: Group A: Subject on study drug (Lovaza) and not on Aspirin, Clopidogrel, or Warfarin. Subject on escalating doses of Lovaza over a 24 week period.
- Group B: Subject on Lovaza + Aspirin: Group B: Subject on study drug (Lovaza) plus Aspirin (< or = 35mg)and not on Clopidogrel or Warfarin. Subject on escalating doses of Lovaza over a 24 week period.
- Group C: Subject on Lovaza + Clopidogrel + Aspirin: Group C: Subject on study drug (Lovaza) plus Clopidogrel (75mg) and Aspirin (< or = 325mg, and not on Warfarin. Subject on escalating doses of Lovaza over a 24 week period.
- Group D: Subject on Lovaza + Warfarin + Aspirin: Group D: Subject on study drug (Lovaza) plus Warfarin and Aspirin (< or = 325mg, and not on Clopidogrel. Subject on escalating doses of Lovaza over a 24 week period.
Arm/Group | Group A: Subject on Lovaza Only | Group B: Subject on Lovaza + Aspirin | Group C: Subject on Lovaza + Clopidogrel + Aspirin | Group D: Subject on Lovaza + Warfarin + Aspirin
Number analyzed (Participants) | 10 | 7 | 10 | 6
percent
  Baseline (Week 0) | 79.5 [36 to 100] | 0 [0 to 49] | 5.5 [2 to 10] | 8 [2 to 27]
  1 gram Lovaza Daily (Week 6) | 79.5 [73 to 100] | 3 [0 to 8] | 6.5 [2 to 15] | 9 [3 to 58]
  2 grams Lovaza Daily (Week 12) | 87.5 [35 to 93] | 2.5 [0 to 7] | 6 [3 to 10] | 12 [7 to 24]
  4 grams Lovaza Daily (Week 18) | 82 [47 to 82] | 0 [0 to 2] | 4 [2 to 8] | 10 [6 to 18]
  8 grams Lovaza Daily (Week 24) | 83 [80 to 85] | 3 [0 to 85] | 5 [1 to 14] | 22 [14 to 45]

2. Secondary Outcome: The Occurence of Any Type of Bleeding
Description: was there any bleeding occurance during the accessed interval
Time Frame: up to and including closeout at 24 weeks
Population: Subjects would indicate if they had any bleeding episode during the trial at each of their testing intervals
Measure: Number; unit: Number of occurance
Arm/Group | Group A: Subject on Lovaza Only | Group B: Subject on Lovaza + Aspirin | Group C: Subject on Lovaza + Clopidogrel + Aspirin | Group D: Subject on Lovaza + Warfarin + Aspirin
Number analyzed (Participants) | 10 | 12 | 10 | 11
Number of occurance | 0 | 1 | 0 | 0

3. Primary Outcome: Bleeding Time
Description: Bleeding time is a measure of how well platelets interact with blood vessel walls to form a clot. A manual blood pressure cuff is placed 2 inches above the antecubital fossa and inflated to 40mmHg. Using a standard Surgicutt device, a small incision is made and a stopwatch is started. The incision edge is blotted at 30 second intervals with standard filter paper until the bleeding has stopped. The time to hemostasis is noted.
Time Frame: up to and including closeout at 24 weeks
Population: Based on number of subjects completing 24 weeks
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Group A: Subject on Lovaza Only | Group B: Subject on Lovaza + Aspirin | Group C: Subject on Lovaza + Clopidogrel + Aspirin | Group D: Subject on Lovaza + Warfarin + Aspirin
Number analyzed (Participants) | 10 | 7 | 10 | 6
seconds
  Baseline (Week 0) | 150 [120 to 180] | 240 [210 to 330] | 570 [440 to 720] | 240 [195 to 330]
  1 gram Lovaza Daily (Week 6) | 240 [180 to 300] | 345 [240 to 450] | 720 [450 to 720] | 285 [218 to 323]
  2 grams Lovaza Daily (Week 12) | 240 [180 to 270] | 390 [330 to 450] | 690 [540 to 720] | 285 [188 to 330]
  4 grams Lovaza Daily (Week 18) | 255 [180 to 270] | 330 [300 to 420] | 600 [360 to 780] | 240 [210 to 300]
  8 grams Lovaza Daily (Week 24) | 255 [210 to 300] | 360 [330 to 420] | 600 [60 to 720] | 270 [195 to 323]
Statistical Analysis 1: Comparison: Group B: Subject on Lovaza + Aspirin; Group B baseline vs. Group B Week 12; Test type: Superiority or Other; p = 0.01, Wilcoxon (Mann-Whitney) — A P-value <0.05 when compared to baseline is considered significant

4. Primary Outcome: EQELS (Electrophoretic Quasi Elastic Light Scattering: Change in Mobility After the Addition of Arachidonic Acid
Description: Measurements were made using a modified device (EQELS) to specifications of constant current, high electric field and a scattering angle of 30 degrees. EQELS provides a sensitive assessment of subtle changes in the cell surface that occurs with activation, ligand binding or apoptosis. These changes are the result of different distributions of charged groups that define a surface charge finger print for the current state of activation of the cell. Resting state platelets have a negative surface charge, whereas fully activated platelets have a positive surface charge.
Time Frame: up to and including closeout at 24 weeks
Population: Based on number of subjects completing 24 weeks. Change in EQELS value after the addition of Arachidonic Acid.
Measure: Median (Inter-Quartile Range); unit: mobility units
Arm/Group | Group A: Subject on Lovaza Only | Group B: Subject on Lovaza + Aspirin | Group C: Subject on Lovaza + Clopidogrel + Aspirin | Group D: Subject on Lovaza + Warfarin + Aspirin
Number analyzed (Participants) | 10 | 7 | 10 | 6
mobility units
  Baseline (Week 0) | 0.28 [-0.08 to 1.85] | -0.04 [-1.38 to 0.39] | -1.04 [-1.26 to -0.89] | -1.10 [-1.19 to -0.03]
  1 gram Lovaza Daily (Week 6) | -0.45 [-0.93 to 0.18] | -0.72 [-1.03 to -0.37] | -0.73 [-1.09 to 0.56] | -0.50 [-0.79 to 0.09]
  2 grams Lovaza Daily (Week 12) | -0.95 [-1.11 to -0.55] | -1.30 [-1.62 to -1.17] | -1.29 [-1.40 to -1.05] | -0.58 [-1.01 to 0.27]
  4 grams Lovaza Daily (Week 18) | -1.08 [-1.39 to -0.99] | -0.94 [-1.11 to -0.89] | -1.14 [-1.29 to -0.94] | -0.44 [-1.91 to 0.76]
  8 grams Lovaza Daily (Week 24) | -0.88 [-1.15 to -0.80] | -0.97 [-1.09 to -0.83] | -0.89 [-1.31 to -0.80] | -0.19 [-0.76 to 0.26]
Statistical Analysis 1: Comparison: Group A: Subject on Lovaza Only vs Group B: Subject on Lovaza + Aspirin vs Group C: Subject on Lovaza + Clopidogrel + Aspirin; The median of Groups A, B, and C grouped together was compared Baseline to Week 6; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Group A: Subject on Lovaza Only vs Group B: Subject on Lovaza + Aspirin vs Group C: Subject on Lovaza + Clopidogrel + Aspirin; The median of Groups A, B, and C grouped together was compared Baseline to Week 12; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: Each patient was monitored for the full time period of 24 weeks, unless withdrawn from study early.
Groups:
- Group A: Lovaza only
- Group B: Lovaza plus aspirin
- Group C: Lovaza plus clopidogrel
- Group D: Lovaza plus aspirin plus coumadin
Arm/Group | Group A | Group B | Group C | Group D
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/12 | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 4/12 | 0/10 | 2/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=10) | Group B (N=12) | Group C (N=10) | Group D (N=11)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Attributed to drug (intervention). Discontinued the study prior to Week 24 (Week 20, Week 21).
GI problem (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Attributed to drug (intervention). Discontinued the study prior to Week 24 (Week 14, Week 18).
Minor Bleeding (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject had finger injury with minor bleeding that was a concern. The subject withdrew from study at 12 week testing interval.
Elevated liver enzymes (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Subject was removed from study by physician.
Unknown medical issue (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Subject was withdrawn from study at 18 Week testing period due to undefined medical issue.

LIMITATIONS AND CAVEATS:
Major limitation for this pilot study was the small number of patients analyzed per group. Despite the small numbers we were able to show the statistical significance for a change in the platelet surface charge with Lovaza.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No